CLINICAL TRIAL: NCT06454994
Title: A Prospective, Multicentric, Comparative, Split-face Clinical Study to Evaluate Safety and Effectiveness of Noble Lift® Lifting Threads
Brief Title: Clinical Study to Evaluate Safety and Effectiveness of Noble Lift® Lifting Threads
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Co., Ltd (Industry)
Collaborators: Eurofins Laboratoire Dermscan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 23E1359
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Aesthetic
Keywords: Lifting threads; Eyebrow lift; Jaw laxity

STUDY DESIGN:
Intervention Model Description: Hemi-face, intra-individual study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noble Lift threads (Experimental)
  Interventions: Device: Eyebrow lift; Device: Jaw lift
- Croquis threads (Active Comparator)
  Interventions: Device: Eyebrow lift; Device: Jaw lift

INTERVENTIONS:
Device: Eyebrow lift — Upper face lifting
Device: Jaw lift — Mid-face and low-face lifting

SUMMARY:
The aim of this study is to compare two models of the Nobel Lift range (PDO sutures) with similar PDO devices available on the market, in a split-face comparative study. Each thread model will be used in one indication: upper face (eyebrow lift) or mid-face and lower-face.

Aesthetic efficacy of the devices will be evaluated and compared with the Global Aesthetic Improvement Scale (GAIS), jowl laxity scale, subjective evaluation of the patient and photographs during a 12-months period. Safety of the devices and procedures will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* BMI comprised between 18.5 and 30
* No ongoing or planned diet.
* Group 1: requiring an aesthetic treatment of upper face with resorbable threads.
* Group 2: Subject requiring an aesthetic treatment of mid-face and lower-face with resorbable threads
* Subject with dense and not too thin skin.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study;
* Suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study result and/or subject safety, especially cardiac disorder, non-controlled high blood pressure, diabetes, panic disorders, depression, active auto-immune disease, cold, high fever,…
* Suffering from malnutrition.
* Acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.
* Wound healing disorder or with a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
* History of precancerous lesions/skin malignancies.
* Active skin disease within 6 months of study entry.
* Scars, rosacea, herpes, acne, blotches or other pathology in the face, at the investigator appreciation.
* Predisposed to keloidosis or hypertrophic scarring.
* Known history of hyper- or hypo-pigmentation in the face.
* Known history of multiple allergies, allergic/anaphylactic reactions including allergy/ hypersensitivity to lidocaine, anaesthetics of the amide type, the used antiseptic components, the used antibiotic cream components.
* Known bleeding disorder or is receiving medication that will likely increase the risk of bleeding during treatment.
* Extensive skin laxity, thin skin and/or severe malar fat sagging.
* Foreign body sensitivity or known or suspected allergies to implant or instrument materials in particular plastic/biomaterial.
* Any medication which may interfere, at the interpretation of the investigator, with the study objectives in term of efficacy and safety/tolerance.
* Dental care in the past 2 weeks or who planned to receive dental care in the 2 months after the treatment.
* Anticoagulant (such as aspirin, warfarin, blood circulation enhancer and clotbuster) during the week before the injection session .
* Chemotherapy agents, immunosuppressive medications or systemic corticosteroids in the past 3 months and during the study.
* Lifting of the face in the past 12 months or other surgery of the face in the past 6 months.
* Resorbable fillers within the past 12 months, other resorbable threads within the past 12 months, neurotoxin in the past 5 months or plans to receive such treatments during the study.
* Permanent filler on the face.
* Subcutaneous permanent retaining structure on the face (meshing, permanent threads, gold strand etc.).
* Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Global Aesthetic Improvement (GAIS) by the investigator between both products | Month 3
  Non-inferiority of Noble Lift® threads in comparison with Croquis® thread, in terms of GAIS mean score on Month 3, assessed by an independent blinded investigator on photos (in global and for each indication). GAIS is a scale from 1 (worse) to 5 (very much improved).

SECONDARY OUTCOMES:
Percentages of responders for Global Aesthetic Improvement (GAIS) by the investigator | Month 3, Month 6, Month 12
  GAIS is a scale from 1 (worse) to 5 (very much improved)
Percentages of responders for Global Aesthetic Improvement (GAIS) by the subject | Month 3, Month 6, Month 12
  GAIS is a scale from 1 (worse) to 5 (very much improved)
Change from baseline of Facial Laxity Rating Scale (FLRS) score | Month 3, Month 6, Month 12
  FLRS is a scale from 1 (mild laxity) to 9 (severe laxity)
Percentages of subjects satisfied with the intervention using a subjective evaluation questionnaire | Month 3, Month 6, Month 12
  Answers are evaluated from 1 (very dissatisfied) to 5 (very satisfied)
Number and percentages of immediate and early skin reactions collected by the subject | Month 1
  Skin reactions are scored as mild, moderate or severe
Number and percentages of skin reactions scored by the investigator | Month1, Month 3, Month 6, Month 12
  Skin reactions are scored as mild, moderate or severe
Number and percentages of Adverse Events | Month1, Month 3, Month 6, Month 12

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Dr Jeanblanc, Aix-en-Provence
  - Dr Facchinetti, Cannes
  - Dr Converset-Viethel, Lyon
  - Dr Lemmel, Paris

IPD SHARING:
Plan to Share IPD: No